CLINICAL TRIAL: NCT05315544
Title: CSI Percutaneous Ventricular Assist Device (pVAD) First in Human Study
Brief Title: Cardiovascular Systems Inc. (CSI) pVAD First in Human Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN-0015-P
Record Dates: First submitted 2022-03-26; First posted 2022-04-07 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
Keywords: pVAD; High risk PCI; Cardiovascular Systems, Inc.; Mechanical Circulatory Support (MCS)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CSI pVAD (Experimental)
  Interventions: Device: CSI pVAD system

INTERVENTIONS:
Device: CSI pVAD system — The CSI percutaneous ventricular assist device (pVAD) is being investigated as a temporary left ventricular system intended to support and/or provide hemodynamic stability during high-risk percutaneous coronary interventions.

SUMMARY:
This study will collect initial clinical data on the CSI pVAD system to inform device design and finalization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non- pregnant female ≥ 18 years of age
2. Life expectancy ≥ 1 year
3. Ejection Fraction (EF) >15% and ≤ 40%
4. Scheduled for an elective high risk percutaneous coronary intervention

Exclusion Criteria:

1. Hemodynamically unstable MI with elevated cardiac biomarker and no evidence of at least 1 consecutive CK-MB or troponin value trending downward from a previous value OR ST-Elevation Myocardial Infarction (STEMI) within 14 days of Index Procedure
2. Pre-Procedure cardiac arrest within 24 hours of enrollment requiring cardiopulmonary resuscitation
3. Cardiogenic shock
4. Left ventricular (LV) mural thrombus
5. Presence of a prosthetic valve or a heart constrictive device
6. Aortic stenosis
7. Moderate or severe aortic regurgitation (≥ 2+ by echo)
8. Severe peripheral vascular disease that will preclude the use of a 12F access sheath, which is required for the insertion of the CSI pVAD catheter
9. Severe aortic tortuosity
10. Severe aortic calcification
11. Vasculature will not tolerate a right heart catheterization
12. Renal dysfunction (serum creatinine ≥ 2.5 mg/dl) or requirement for hemodialysis
13. Liver dysfunction with elevation of liver enzymes and bilirubin levels to ≥ 3X upper lab normal (ULN) or Internationalized Normalized Ratio (INR) ≥ 2 or lactate dehydrogenase (LDH) > 2.5X ULN
14. Uncorrectable abnormal coagulation parameters
15. History of heparin induced thrombocytopenia
16. Sustained ventricular tachycardia
17. Stroke or transient ischemic attack (TIA) within 6 months or any permanent neurological deficit
18. Chronic anemia (hemoglobin < 8 g/dL)
19. Subject may require long term support with a commercially available hemodynamic support device
20. Active systemic infection requiring oral or intravenous antibiotics
21. Allergy or intolerance to ionic and nonionic contrast media, anticoagulants, or antiplatelet therapy drugs that cannot be adequately premedicated
22. Allergy or intolerance to system components
23. Participation in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Procedural success | Intraprocedural
  Delivery of the device to the correct anatomical position, successful operation and removal of the CSI pVAD system
Intraprocedural Major Device-Related Adverse Events | 24-hours Post-Index Procedure
  Composite incidence of:
  * Cardiovascular death
  * Clinically significant myocardial infarction (MI) defined as the composite of MI events per Society for Cardiovascular Angiography and Intervention (SCAI) periprocedural MI and Fourth Universal MI definitions
  * Any repeat revascularization (PCI or CABG)
  * Stroke defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Chambers, MD, Study Director — Abbott Medical Devices
Locations (1):
- Tbilisi Heart & Vascular, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No